CLINICAL TRIAL: NCT04074915
Title: Effects of 1% Matricaria Chamomile Mouth Rinse for the Management of Chronic Periodontitis: a Double Blind Randomized, Placebo Controlled Clinical Trial
Brief Title: Effects of Herbal Mouth Rinse for Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Dental Sciences, Bareilly, Uttar Pradesh, India (Other)
Responsible Party: Principal Investigator, ASHISH AGARWAL, Clinical professor, institute of dental sciences, bareilly, Institute of Dental Sciences, Bareilly, Uttar Pradesh, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEC/IDS/38/2019
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo rinse (Placebo Comparator): Normal saline
  Interventions: Other: Placebo mouth rinse
- Chlorhexidine mouth rinse (Experimental): Chlorhexidine mouth rinse
  Interventions: Drug: Chlorhexidine mouth rinse
- Test group (Experimental): Chamomile mouth rinse
  Interventions: Drug: Test group

INTERVENTIONS:
Other: Placebo mouth rinse — Normal saline
  Other Names: NS
  Arms: Placebo rinse
Drug: Chlorhexidine mouth rinse — Chlorhexidine gluconate
  Other Names: CHX
  Arms: Chlorhexidine mouth rinse
Drug: Test group — Chamomile mouth rinse
  Other Names: CMT
  Arms: Test group

SUMMARY:
This double blind, randomized, placebo controlled, parallel clinical trial involved seventy five patients, suffering with chronic periodontitis, which were randomly divided in three groups: negative control (SRP+placebo), positive control (SRP+0.12% CHX), and test group (SRP+1% MTC mouth rinse). Mouth rinsing (adjunctive therapy) was continued for 1 month while clinical parameters [plaque index (PI), gingival index (GI), sulcus bleeding index (SBI), probing pocket depth (PPD), clinical attachment level (CAL), gingival recession (GR), stain index (SI)] were evaluated at base line, 1 month, and 3 months. CFU was also evaluating at above said time periods.

DETAILED DESCRIPTION:
This double blind, randomized, placebo controlled, parallel clinical trial involved seventy five patients, suffering with chronic periodontitis, which were randomly divided in three groups: negative control (SRP+placebo), positive control (SRP+0.12% CHX), and test group (SRP+1% MTC mouth rinse). Mouth rinsing (adjunctive therapy) was continued for 1 month.The primary outcome of this study was CAL, while PPD was the secondary outcome measure. A single clinician (AA) who was blinded to the groups assigned to the individuals, recorded all the parameters i.e. PI, GI, SBI, PPD, CAL, GR, SI at base line (prior to the treatment), 1 and 3 months after therapy. PPD, CAL and GR were recorded at the six sites per tooth in every tooth, except third molar, with a manual UNC-15 periodontal probe (Hu-Friedy, Leinmen, Germany) to the nearest millimeter. For recording of parameters at different time periods patients were instructed to refrain from any oral hygiene procedure for 8 hours prior to the evaluation. Staining of the six maxillary anterior teeth was assessed using the Lobene index. CFUs of P. ginigvalis, T. forsythia, and T. denticola were evaluated at baseline , 1 months, 3 months.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy individuals of > 30 years of age with previously untreated generalized chronic periodontitis (defined by Armitage in 1999),
* having minimum 15 teeth,
* minimum of six teeth with at least one interproximal site with PPD between 5-7mm,
* CAL between 5-10 mm, at least 30% of the sites with PPD and CAL ≥ 5 mm
* presence of bleeding on probing (BOP).

Exclusion Criteria:

* was any systemic disease,
* use of any medication in the previous 6 months,
* subjects wearing partial removal prosthesis or orthodontic appliance,
* allergy to ingredient used in the study, alcoholics, smokers or tobacoo users in any form, mentally retarded individual, pregnant or lactating females.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Clinical attachment loss | 3 Months
  Distance from cemento enamel junction to base of the pocket

SECONDARY OUTCOMES:
Probing pocket depth | 3 Months
  Distance from ginigval margin to base of the pocket
colony forming units | 3 months
  numbers of colonies of bacteria using anaerobic culture

CONTACTS AND LOCATIONS:
Locations (1):
- Ashish Agarwal, Bareilly, Uttar Pradesh, India